CLINICAL TRIAL: NCT00692237
Title: Cardiovascular Effects of Chronic Sildenafil (Viagra) Treatment in Diabetic Subjects With Endothelial Dysfunction.
Brief Title: Cardiovascular Effects of Chronic Sildenafil in Men With Type 2 Diabetes
Acronym: CECSID
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Andrea M. Isidori, Professor, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 746/07
Record Dates: First submitted 2008-06-04; First posted 2008-06-06 (Estimated); Results first posted 2012-05-15 (Estimated); Last update posted 2013-05-08 (Estimated); Status verified 2013-05

CONDITIONS: Diabetes Mellitus, Type 2; Endothelial Dysfunction
Keywords: Type 2 diabetes mellitus; Endothelial dysfunction; Sildenafil
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sildenafil Citrate

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Sildenafil 100 mg
  Interventions: Drug: Sildenafil
- 2 (Placebo Comparator): Placebo 100 mg
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sildenafil — 100 mg daily (3 capsules/day)
  Other Names: - Viagra 25 mg; - Viagra 50 mg
  Arms: 1
Drug: Placebo — Placebo 100 mg (3 capsules/day)
  Arms: 2

SUMMARY:
Type 2 Diabetes Mellitus (T2DM) represents a model of endothelial dysfunction, where chronic nitric oxide deprivation, hyperglycaemia and hyperinsulinemia and fibrogenic mediators lead to cardiovascular remodelling associated with diabetic cardiomyopathy and in consequence to secondary complications of diabetes. Specific anti-oxidative and anti-fibrotic therapies are not currently available. Sildenafil (Viagra) has demonstrated the capability of significantly improving endothelial dysfunction and cardiac fibrosis in experimental animal models.

The purpose of the present study is performed to establish the effect of chronic high dose sildenafil treatment on heart performance in diabetic subjects.

DETAILED DESCRIPTION:
Type 2 Diabetes Mellitus (T2DM) represents a model of endothelial dysfunction at central and peripheral levels, where chronic nitric oxide deprivation, due to hyperglycaemia, leads to a loss of vascular endothelium-relaxant function and ischaemia-reperfusion ventricular damage. Since haemodynamic and oxidative stress could trigger a pro-inflammatory process of the intracardiac vasculature, endothelial cells activated in turns can produce fibrogenic mediators and induce fibroblast activation and myocardial fibrosis. Moreover, the increase of insulin levels of T2DM induces cardiotoxicity increasing the expression of ventricular angiotensin II type 1 receptor (AT1). All these mechanisms lead to cardiovascular remodelling associated with diabetic cardiomyopathy that is characterized by an impairment of heart diastolic performance with a ventricular hypertrophy and a dilatation and an increase of heart torsion.

Specific anti-oxidative and anti-fibrotic therapies are not currently available. Phosphodiesterase 5 inhibitors (PDE5i) work to improve endothelial dysfunction by preventing the breakdown of cyclic guanosine monophosphate (cGMP), resulting in increased cellular content and consequent relaxation of smooth muscle cells of all systemic arteries and veins. PDE5i have therefore the potential to impact the cardiovascular performance, acting on all these mechanisms.

The aim of the study is to evaluate the cardiovascular effects of the chronic (3 months) high dose (100 mg daily) sildenafil treatment in patient with type 2 diabetes. We will analyze the changes in parameters of endothelial dysfunction and heart remodelling and in metabolic indices. We will evaluate the outcomes at day 90. Moreover we will estimate if the changes in endothelial function will be sustained 30 days after discontinuing treatment.

This is designed as a phase IV study on chronic treatment with a cohort size of 30 patients randomized to receive Sildenafil and 20 patients randomized to placebo. Accounting for a 15% drop off, a total enrollment of 60 patients is planned. Patients will begin a washout from PDE5i in the first visit (4 weeks before the beginning of the treatment). Evaluation of potential toxicity will be monitored throughout the course of treatment. Follow-up visits will take place at days + 30, +60, +90 (end of treatment) and +120. Plasma and serum monitoring of basal and postprandial glycaemia and insulinemia, hematochemical routine, VEGF, hormones and others cytokines and albuminuria will be made prior to treatment, at days 30, 60, 90, 120. Measurements of cine-MRI, FMD and blood pressure Holter 24h will be made at time 0 and at days 90.

The long-term objective is to identify a safe and easily administered treatment that improves functional outcome in diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 2 diabetes mellitus
* Patients age 35-75
* Metabolic control of diabetes by diet or oral treatment (unmodified in the last 3 months)
* Blood pressure <160/100 mmHg, including subjects with controlled hypertension, treated with ACE-inhibitors/sartans, unmodified in the last 3 months

Exclusion Criteria:

* Participation in another study with an investigational drug or device
* HbA1c >12%
* Alterations during ECG stress examination
* Current use of nitrate agents
* Proliferative retinopathy
* Patients with history of cardiovascular and malignant disease
* Psychosocial disturbance
* Alcohol or drug dependence
* Allergy or hypersensitivity to sildenafil or other Phosphodiesterase inhibitors.

Ages: 35 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2008-01; Primary Completion 2009-09 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Lenzi, MD, PhD, Principal Investigator — University of Roma La Sapienza
Locations (1):
- Dipartimento di Fisiopatologia Medica - Policlinico Umberto I, Rome, Italy

REFERENCES:
- [Result] Giannetta E, Isidori AM, Galea N, Carbone I, Mandosi E, Vizza CD, Naro F, Morano S, Fedele F, Lenzi A. Chronic Inhibition of cGMP phosphodiesterase 5A improves diabetic cardiomyopathy: a randomized, controlled clinical trial using magnetic resonance imaging with myocardial tagging. Circulation. 2012 May 15;125(19):2323-33. doi: 10.1161/CIRCULATIONAHA.111.063412. Epub 2012 Apr 11. PMID 22496161
- [Derived] Pofi R, Giannetta E, Galea N, Francone M, Campolo F, Barbagallo F, Gianfrilli D, Venneri MA, Filardi T, Cristini C, Antonini G, Badagliacca R, Frati G, Lenzi A, Carbone I, Isidori AM. Diabetic Cardiomiopathy Progression is Triggered by miR122-5p and Involves Extracellular Matrix: A 5-Year Prospective Study. JACC Cardiovasc Imaging. 2021 Jun;14(6):1130-1142. doi: 10.1016/j.jcmg.2020.10.009. Epub 2020 Nov 18. PMID 33221242
- [Derived] Venneri MA, Barbagallo F, Fiore D, De Gaetano R, Giannetta E, Sbardella E, Pozza C, Campolo F, Naro F, Lenzi A, Isidori AM. PDE5 Inhibition Stimulates Tie2-Expressing Monocytes and Angiopoietin-1 Restoring Angiogenic Homeostasis in Diabetes. J Clin Endocrinol Metab. 2019 Jul 1;104(7):2623-2636. doi: 10.1210/jc.2018-02525. PMID 31102457
- [Derived] Mandosi E, Giannetta E, Filardi T, Lococo M, Bertolini C, Fallarino M, Gianfrilli D, Venneri MA, Lenti L, Lenzi A, Morano S. Endothelial dysfunction markers as a therapeutic target for Sildenafil treatment and effects on metabolic control in type 2 diabetes. Expert Opin Ther Targets. 2015;19(12):1617-22. doi: 10.1517/14728222.2015.1066337. Epub 2015 Jul 15. PMID 26178526

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible men were recruited from the outpatient clinics of Policlinico Umberto I - Sapienza University Hospital of Rome between 2008 and 2009.
Pre-assignment Details: Overall 66 patients were eligible and enrolled; Seven were then excluded due to evidence of aneurysm of ascending aorta (1) on stress-Echo and of ischemic heart disease (6) at the first CMR. Fifty-nine patients were randomized.
Groups:
- Sildenafil: Sildenafil citrate 100 mg/day (50+25+25)
- Placebo: Placebo 100 mg/day (50 + 25 + 25)
Period: Overall Study
Arm/Group | Sildenafil | Placebo
Started | 30 | 29
Completed | 29 | 25
Not Completed | 1 | 4
Not completed — Withdrawal by Subject | 1 | 3
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sildenafil | Placebo | Total
Number analyzed (Participants) | 30 | 29 | 59
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 20 | 40
  >=65 years | 10 | 9 | 19
Age Continuous [Mean (Standard Deviation); unit: years] | 61 (7) | 59 (7) | 60 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 30 | 29 | 59
Region of Enrollment [Number; unit: participants]
  Italy | 30 | 29 | 59

OUTCOME MEASURES:

1. Primary Outcome: Left Ventricular Torsion Defined as Change in Ventricular Mid-wall Rotation (°) Measured by Cine-Cardiac Magnetic Resonance (CMR) Imaging With Tagging, Before and After Three Months of Treatment With Sildenafil and Placebo (100 mg/Day).
Description: Diabetic cardiomyopathy and hypertrophy are characterized by an increase in cardiac torsion Normal value of rotation are < 12°; in hypertrophic heart such values can raise up to 20-25°. A reduction in left ventricular wall rotation is a sign of improvement after removal of known causes of hypertrophy (for example after surgical repair of aortic stenosis). Based on previous studies a reduction of 3 degrees (°) is considered clinically significant.
Time Frame: 0 and + 3 months
Population: An overall sample size of 32 subjects (16 for each group) would thus have given a 90% power to detect the specified minimum detectable difference (3°) at a 2-sided significance level of 0.01; 59 patients were enrolled: 29 randomized to Sildenafil and 25 randomized to Placebo completed the trial. Analysis was per primary efficacy outcome (LV-q).
Measure: Mean (Standard Deviation); unit: Degree angle (delta)
Groups:
- Sildenafil: Patients randomized to receive sildenafil were instructed to take 3 capsules per day (25 mg at 8.00 a.m. + 25 mg at 4.00 p.m. + 50 mg at 10.00 p.m.) that were identical-looking to placebo capsules, for a duration of 3 months (12 weeks). The allocation list was produced using dedicated software by permuted-block randomization with 1:1 allocation using randomly sized blocks (4 to 8). The study was double-blinded.
- Placebo: Patients randomized to receive placebo were instructed to take 3 capsules per day (1 at 8.00 a.m. + 1 at 4.00 p.m. + 1 at 10.00 p.m.) that were identical-looking to sildenafil capsules, for a duration of 3 months (12 weeks). The allocation list was produced using dedicated software by permuted-block randomization with 1:1 allocation using randomly sized blocks (4 to 8). The study was double-blinded.
Arm/Group | Sildenafil | Placebo
Number analyzed (Participants) | 29 | 25
Degree angle (delta) | -3.89 (3.11) | 2.13 (2.35)

2. Secondary Outcome: Ejection Fraction (EF) Defined as the Volume of Blood Ejected With Each Beat Was Measured on Cine-Cardiac Magnetic Resonance (CMR) Images Before and After Three Months Treatment With Sildenafil and Placebo (100 mg/Day).
Description: The volume of blood within a ventricle immediately before a contraction is known as the end-diastolic volume; the volume of blood left in a ventricle at the end of contraction is end-systolic volume. The difference between end-diastolic volume and end-systolic volumes is the volume of blood ejected with each beat. Ejection fraction (Ef) is the fraction of the end-diastolic volume that is ejected with each beat; expressed as percentage of EDV. This is a measure of cardiac performance that can be deteriorated in diabetic cardiomyopathy.
Time Frame: 0 and + 3 months
Population: We included in this analysis all the patients that concluded the study (Sildenafil group = 29; Placebo group = 25).
  The 4 randomized patients who discontinued, did not perform the second after-treatment CMR evaluation.
  Analysis was "per protocol".
Measure: Mean (Standard Deviation); unit: Percentage % of volume (delta)
Arm/Group | Sildenafil | Placebo
Number analyzed (Participants) | 29 | 25
Percentage % of volume (delta) | 2.77 (4.36) | 3.14 (5.87)

ADVERSE EVENTS:
Arm/Group | Sildenafil | Placebo
Serious Adverse Events (participants affected / at risk) | 0/30 | 1/29
Other Adverse Events (participants affected / at risk) | 0/30 | 0/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sildenafil (N=30) | Placebo (N=29)
Portal Vein Thrombosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes